CLINICAL TRIAL: NCT05449080
Title: Disorders of Sex Development (DSD) 46.XY Due to Type 2 5-Α Reductase Deficiency in Three Siblings: Case Report From a Low-Resource Setting
Brief Title: Disorders of Sex Development (DSD) 46.XY in Three Siblings
Status: Completed | Type: Observational
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Other Study IDs: OBGY-202206.03
Record Dates: First submitted 2022-06-26; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Genotype
Keywords: Disorders of Sex Development; Type 2 5-alpha reductase deficiency
MeSH Terms: conditions — Disorders of Sex Development | interventions — Karyotype

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: subjects with type 2 5-alpha reductase deficiency
  Interventions: Diagnostic Test: Karyotype

INTERVENTIONS:
Diagnostic Test: Karyotype — Patients were subjected to karyotype to determine their genotype

SUMMARY:
This is a case series of three siblings with DSD 46,XY with relevant discussion

DETAILED DESCRIPTION:
This is a case series of three sisters with DSD 46 X,Y. Three sisters, aged nineteen, seventeen, and fifteen years old came with an identical complaint of late menarche. Physical examinations, lab results and karyotypes were performed.

ELIGIBILITY:
Inclusion Criteria:

* 3 female siblings with identical complaints of no menarche

Exclusion Criteria:

* patients outside this family.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients were 3 female siblings with identical complaints of no menarche of varying ages. Patients were subjected to physical examination, lab tests and karyotype to determine their genotypes.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Karyotype | 1 month after testing
  Patient's karyotype

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Universitas Padjadjaran, Bandung, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
Anonymous data on female subjects may be shared with reasonable written request to the authors.

REFERENCES:
- [Background] Marzuki NS, Idris FP, Kartapradja HD, Harahap AR, Batubara JRL. Characterising SRD5A2 Gene Variants in 37 Indonesian Patients with 5-Alpha-Reductase Type 2 Deficiency. Int J Endocrinol. 2019 Dec 1;2019:7676341. doi: 10.1155/2019/7676341. eCollection 2019. PMID 31885560
- [Result] Walter KN, Kienzle FB, Frankenschmidt A, Hiort O, Wudy SA, van der Werf-Grohmann N, Superti-Furga A, Schwab KO. Difficulties in diagnosis and treatment of 5alpha-reductase type 2 deficiency in a newborn with 46,XY DSD. Horm Res Paediatr. 2010;74(1):67-71. doi: 10.1159/000313372. Epub 2010 Apr 16. PMID 20395661